CLINICAL TRIAL: NCT04524871
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Advanced Liver Cancers (Morpheus-Liver)
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Advanced Liver Cancers (Morpheus-Liver)
Acronym: MORPHEUS-LIVER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Adagene Inc (Industry); Tempest Therapeutics (Industry); NiKang Therapeutics, Inc. (Industry); Immune-Onc Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42216
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Liver Cancers
MeSH Terms: interventions — atezolizumab; Bevacizumab; Tiragolumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Stage 1: Atezolizumab + Bevacizumab (Active Comparator): Participants will receive atezolizumab plus bevacizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg
- Stage 1: Atezolizumab + Bevacizumab + Tiragolumab (Experimental): Participants will receive atezolizumab plus bevacizumab plus tiragolumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: Tiragolumab
- Stage 1: Atezolizumab + Bevacizumab + Tocilizumab (Experimental): Participants will receive atezolizumab plus bevacizumab plus tocilizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: Tocilizumab
- Stage 1: Atezolizumab + Bevacizumab + TPST-1120 (Experimental): Participants will receive atezolizumab plus bevacizumab plus TPST-1120 until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: TPST-1120
- Stage 1: Tobemstomig 2100 mg Q2W + Bevacizumab (Experimental): Participants will receive Tobemstomig plus bevacizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Bevacizumab 15 mg/kg; Drug: Tobemstomig 2100 mg; Drug: Bevacizumab 10 mg/kg
- Stage 1: Tobemstomig 600 mg Q3W + Bevacizumab (Experimental): Participants will receive Tobemstomig plus bevacizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Bevacizumab 15 mg/kg; Drug: Tobemstomig 600 mg
- Stage 1: Tobemstomig 1200 mg Q3W + Bevacizumab (Experimental): Participants will receive Tobemstomig plus bevacizumab until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Bevacizumab 15 mg/kg; Drug: Tobemstomig 1200 mg
- Stage 1: Atezolizumab + Bevacizumab + ADG126 (Experimental): Participants will receive atezolizumab plus bevacizumab plus ADG126 until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: ADG126
- Stage 1: Atezolizumab + Bevacizumab + IO-108 1200 mg Q3W (Experimental): Participants will receive atezolizumab plus bevacizumab plus IO-108 until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: IO-108 1200 mg
- Stage 1: Atezolizumab + Bevacizumab + NKT2152 (Experimental): Participants will receive atezolizumab plus bevacizumab plus NKT2152 until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab 15 mg/kg; Drug: NKT2152
- Stage 1: Atezolizumab + Bevacizumab+ IO-108 1800 mg Q3W (Experimental): Participants will receive atezolizumab plus bevacizumab plus IO-108 until unacceptable toxicity or loss of clinical benefit, as determined by the investigator after an integrated assessment of radiographic andbiochemical data, local biopsy results (if available), and clinical status
  Interventions: Drug: IO-108 1800 mg

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg by IV on Day 1 of each 21 day cycle.
  Other Names: Tecentriq
  Arms: Stage 1: Atezolizumab + Bevacizumab; Stage 1: Atezolizumab + Bevacizumab + ADG126; Stage 1: Atezolizumab + Bevacizumab + IO-108 1200 mg Q3W; Stage 1: Atezolizumab + Bevacizumab + NKT2152; Stage 1: Atezolizumab + Bevacizumab + TPST-1120; Stage 1: Atezolizumab + Bevacizumab + Tiragolumab; Stage 1: Atezolizumab + Bevacizumab + Tocilizumab
Drug: Bevacizumab 15 mg/kg — Bevacizumab will be administered at a dose of 15 mg/kg by IV infusion on Day 1 of each 21 day cycle.
  Other Names: Avastin
  Arms: Stage 1: Atezolizumab + Bevacizumab; Stage 1: Atezolizumab + Bevacizumab + ADG126; Stage 1: Atezolizumab + Bevacizumab + IO-108 1200 mg Q3W; Stage 1: Atezolizumab + Bevacizumab + NKT2152; Stage 1: Atezolizumab + Bevacizumab + TPST-1120; Stage 1: Atezolizumab + Bevacizumab + Tiragolumab; Stage 1: Atezolizumab + Bevacizumab + Tocilizumab; Stage 1: Tobemstomig 1200 mg Q3W + Bevacizumab; Stage 1: Tobemstomig 2100 mg Q2W + Bevacizumab; Stage 1: Tobemstomig 600 mg Q3W + Bevacizumab
Drug: Tiragolumab — Tiragolumab will be administered at a dose of 600 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Stage 1: Atezolizumab + Bevacizumab + Tiragolumab
Drug: Tocilizumab — Tocilizumab will be administered at a dose of 8 mg/kg by IV infusion on Day 1 of each 21 day cycle.
  Other Names: Actemra
  Arms: Stage 1: Atezolizumab + Bevacizumab + Tocilizumab
Drug: TPST-1120 — TPST-1120 will be administered at a dose of 1200 mg by mouth on Days 1-21 of each 21 day cycle.
  Arms: Stage 1: Atezolizumab + Bevacizumab + TPST-1120
Drug: Tobemstomig 2100 mg — Tobemstomig will be administered at a dose of 2100 mg by IV infusion on Days 1 and 15 of each 28 day cycle.
  Arms: Stage 1: Tobemstomig 2100 mg Q2W + Bevacizumab
Drug: Bevacizumab 10 mg/kg — Bevacizumab will be administered at a dose of 10 mg/kg by IV infusion on Days 1 and 15 of each 28 day cycle.
  Other Names: Avastin
  Arms: Stage 1: Tobemstomig 2100 mg Q2W + Bevacizumab
Drug: Tobemstomig 600 mg — Tobemstomig will be administered at a dose of 600 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Stage 1: Tobemstomig 600 mg Q3W + Bevacizumab
Drug: Tobemstomig 1200 mg — Tobemstomig will be administered at a dose of 1200 mg every 3 weeks.
  Arms: Stage 1: Tobemstomig 1200 mg Q3W + Bevacizumab
Drug: ADG126 — ADG126 will be administered at a dose of 6 mg/kg by IV infusion on Day 1 of every other cycle (cycle length = 21 days).
  Arms: Stage 1: Atezolizumab + Bevacizumab + ADG126
Drug: IO-108 1800 mg — IO-108 will be administered at a dose 1800 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Stage 1: Atezolizumab + Bevacizumab+ IO-108 1800 mg Q3W
Drug: NKT2152 — NKT2152 will be administered by mouth.
  Arms: Stage 1: Atezolizumab + Bevacizumab + NKT2152
Drug: IO-108 1200 mg — IO-108 will be administered at a dose 1200 mg by IV infusion on Day 1 of each 21 day cycle.
  Arms: Stage 1: Atezolizumab + Bevacizumab + IO-108 1200 mg Q3W

SUMMARY:
This is a Phase Ib/II, open-label, multicenter, randomized umbrella study in participants with advanced liver cancers. The study is designed with the flexibility to open new treatment arms as new treatments become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, modify the participant population, or introduce additional cohorts of participants with other types of advanced primary liver cancer.

Cohort 1 will enroll participants with locally advanced or metastatic hepatocellular carcinoma (HCC) who have not received prior systemic therapy for their disease. Eligible participants will initially be randomly assigned to one of several treatment arms (Stage 1). Participants who experience loss of clinical benefit or unacceptable toxicity during Stage 1 may be eligible to receive treatment with a different treatment combination (Stage 2). When a Stage 2 treatment combination is available, this will be introduced by amending the protocol.

ELIGIBILITY:
Inclusion Criteria:

Stage 1

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 7 days prior to randomization
* Locally advanced or metastatic and/or unresectable hepatocellular carcinoma (HCC) with diagnosis confirmed by histology/cytology or clinically by American Association for the Study of
* Liver Diseases criteria in cirrhotic patients
* Child-Pugh class A within 7 days prior to randomization
* Disease that is not amenable to curative surgical and/or locoregional therapies
* No prior systemic treatment for HCC
* Life expectancy >= 3 months
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 and/or additional biomarker status via central testing

Stage 1 and Stage 2

* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1
* Adequate hematologic and end-organ function within 7 days prior to initiation of study treatment
* Documented virology status of hepatitis, as confirmed by screening tests for hepatitis B virus - (HBV) and hepatitis C virus (HCV)
* Negative HIV test at screening
* For women of childbearing potential: agreement to remain abstinent or use contraception and for men: agreement to remain abstinent or use contraception, and agreement to refrain from donating sperm

Stage 2

* ECOG Performance Status of 0, 1, or 2
* Ability to initiate Stage 2 treatment within 3 months after experiencing unacceptable toxicity not related to atezolizumab or RO7247669 or loss of clinical benefit as determined by the investigator while receiving Stage 1 treatment
* Availability of a tumor specimen from a biopsy performed upon discontinuation of Stage 1 (if deemed clinically feasible)

NKT2152-Containing Arm:

* Total bilirubin ≤ 1.5 X ULN in the absence of Gilbert's disease (≤ 3.0 X ULN if Gilbert's disease)
* AST/ALT ≤ 2.5 X ULN (≤ 5 X ULN if liver metastases present)

Exclusion Criteria:

Stage 1

* Prior treatment with CD137 agonists or immune checkpoint blockade therapies or inhibitors targeting HIF2a
* Treatment with investigational therapy within 28 days prior to initiation of study
* Treatment with locoregional therapy to liver within 28 days prior to initiation of study, or non-recovery from side effects of any such procedure
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or at high risk for bleeding
* Prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study
* AEs from prior anti-cancer therapy that have not resolved to Grade <= 1 or better, with the exception of alopecia of any grade
* Inadequately controlled hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease
* History of hemoptysis within 1 month prior to initiation of study
* Evidence of bleeding diathesis or significant coagulopathy
* Current or recent use of aspirin (>325 mg/day) or treatment with clopidogrel, dipyramidole, ticlopidine, or cilostazol
* Current or recent use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose
* Core biopsy or other minor surgical procedure within 3 days prior to initiation of study
* History of abdominal or tracheoesophageal fistula, GI perforation, or intra-abdominal abscess, intestinal obstruction and/or clinical signs/symptoms of GI obstruction
* Evidence of abdominal free air not explained by paracentesis or recent surgery
* Serious, non-healing/dehiscing wound, active ulcer, or untreated bone fracture
* Grade >=2 proteinuria
* Metastatic disease involving major airways/blood vessels, or centrally located mediastinal tumor masses of large volume
* History of clinically significant intra-abdominal inflammatory process
* Radiotherapy within 28 days or abdominal/pelvic radiotherapy within 60 days prior to initiation of study with the exception of palliative radiotherapy to bone lesions within 7 days prior to initiation of study
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to initiation of study; or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to initiation of study; or anticipation of need for major surgery during study or non-recovery from side effects of any such procedure
* Chronic daily treatment with NSAID
* Eligible only for control arm

Stage 1 and 2

* Fibrolamellar or sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* History of hepatic encephalopathy
* Moderate or severe ascites
* HBV and HCV coinfection
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of IPF, organizing pneumonia, drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Active TB
* Significant CV disease within 3 months prior to initiation of study, unstable arrhythmia, or unstable angina
* Major surgery, other than for diagnosis, within 4 weeks prior to initiation of study, or anticipated major surgery during study
* History of malignancy other than HCC within 5 years prior to screening
* Severe infection within 4 weeks prior to initiation of study
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients
* Treatment with systemic immunostimulatory, immunosuppressive agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study
* Grade >= 3 hemorrhage or bleeding event within 8 weeks prior to initiation of study treatment
* Patients entering Stage 2: immunotherapy-related adverse events that have not resolved to Grade 1 or better or to baseline at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From randomization until disease progression or loss of clinical benefit (up to approximately 7-9 years)
  ORR, defined as the proportion of participants with a complete response or partial response on two consecutive occasions >=4 weeks apart during Stage 1, as determined by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Randomization to first occurrence of disease progression or death from any cause in Stage 1 (up to approximately 7-9 years)
  PFS after randomization, defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) | Randomization to death from any cause (up to approximately 7-9 years)
  OS after randomization, defined as the time from randomization to death from any cause.
OS at Specific Timepoints | Randomization to a specific timepoint, such as Month 6
  OS at a specific timepoint, such as Month 6
Duration of Response (DOR) | First occurrence of a documented objective response to disease progression or death (up to approximately 7-9 years)
  DOR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1.
Disease Control | Randomization to end of study (approximately 7-9 years)
  Disease control, defined as stable disease for >=12 weeks or a complete or partial response, as determined by the investigator according to RECIST v1.1.
Percentage of Participants With Adverse Events During Stage 1 | Baseline through the end of the study (approximately 7-9 years)
Percentage of Participants With Adverse Events During Stage 2 | Baseline through the end of the study (approximately 7-9 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (16):
  - UC Irvine Medical Center, Costa Mesa, California
  - City of Hope, Duarte, California
  - University of California San Diego, La Jolla, California
  - UC Irvine Medical Center, Orange, California
  - University of California San Francisco Cancer Center, San Francisco, California
  - UCLA Center for East, Santa Monica, California
  - Cherry Creek Medical Center, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - UCHealth Cancer Center Pharmacy - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Parkland Health & Hospital System, Dallas, Texas
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Zhongshan Hospital Fudan University, Shanghai
- France (4):
  - Centre Georges Francois Leclerc, Dijon
  - CHU Hôpitaux de Marseille, Marseille
  - Centre Eugène Marquis, Rennes
  - Gustave Roussy, Villejuif
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah University Medical Center, Jerusalem
  - Davidof Center - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Centre, Tel Aviv
- Auckland City Hospital, Auckland, New Zealand
- South Korea (4):
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Finn RS, Ryoo BY, Hsu CH, Li D, Burgoyne AM, Cotter C, Badhrinarayanan S, Wang Y, Yin A, Edubilli TR, Mahrus S, Secrest MH, Shemesh CS, Yu N, Hack SP, Cha E, Gane E. Tiragolumab in combination with atezolizumab and bevacizumab in patients with unresectable, locally advanced or metastatic hepatocellular carcinoma (MORPHEUS-Liver): a randomised, open-label, phase 1b-2, study. Lancet Oncol. 2025 Feb;26(2):214-226. doi: 10.1016/S1470-2045(24)00679-X. Epub 2025 Jan 21. PMID 39855251